CLINICAL TRIAL: NCT06011759
Title: Maintaining Implementation Through Dynamic Adaptations (MIDAS) - Suicide Prevention 2.0 Clinical Telehealth (SP 2.0) (QUE 20-025)
Brief Title: Maintaining Implementation Through Dynamic Adaptations (MIDAS) Suicide Prevention 2.0 Clinical Telehealth
Acronym: MIDAS SPCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 23-001
Record Dates: First submitted 2023-08-16; First posted 2023-08-25 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Suicidal Self-directed Violence; Suicidal Preparatory Behavior
Keywords: implementation science; implementation strategy; suicide prevention; academic detailing; quality improvement
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: A multi-faceted implementation intervention including qualitative interviews and feedback and optional delivery of Academic Detailing and/or LEAP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): A multi-faceted implementation intervention including qualitative interviews and feedback and optional delivery of Academic Detailing and/or LEAP.
  Interventions: Behavioral: Academic Detailing (AD); Behavioral: LEAP

INTERVENTIONS:
Behavioral: Academic Detailing (AD) — The National Resource Center for Academic Detailing (NaRCAD) describes AD as "an innovative, one-on-one outreach education technique that helps clinicians provide evidence-based care to their patients. Using an accurate, up-to-date synthesis of the best clinical evidence in an engaging format, academic detailers ignite clinician behavior change, ultimately improving patient health. A successful AD visit is highly interactive, always a dialogue, and assesses a clinician's individual needs, beliefs, attitudes, issues, and concerns in order to promote better [practice]."
Behavioral: LEAP — Learn. Engage. Act. Process (LEAP) program is a structured 6-month core curriculum plus 6 monthly collaborative sessions. The LEAP quality improvement program engages frontline teams in sustained incremental improvements of EBPs over a six-month period, allowing space for busy clinicians to learn and immediately apply fundamental QI skills. LEAP encompasses: 1) a structured, accessible curriculum based on the Institute for Healthcare Improvement's (IHI) Model for Improvement and Plan-Do-Study-Act cycles of change; 2) team-based, hands-on learning, and 3) coaching support and a QI network to enhance learning and accountability.

SUMMARY:
Scientific advances are constantly leading to better treatments. However, it is quite challenging for healthcare systems, including VA, to ask very busy providers to change the way they practice. The MIDAS QUERI program helps providers improve the way they treat VA patients. This project will focus on increasing referrals to the Suicide Prevention 2.0 Clinical Telehealth (SP 2.0) initiative through the delivery of Academic Detailing and LEAP (a team-based quality improvement program). SP 2.0 provides accessible, evidence-based suicide prevention treatment to all Veterans with a history of suicidal self-directed violence or preparatory behaviors in the past 12 months.

DETAILED DESCRIPTION:
Sustained integration of evidence-based practices (EBPs) is a challenge within many healthcare systems, especially in settings that have already strived but failed to achieve longer-term goals. The Veterans Affairs (VA) Maintaining Implementation through Dynamic Adaptations (MIDAS) Quality Enhancement Research Initiative (QUERI) program was funded as a series of trials to test multi-component implementation strategies to sustain optimal use of EBPs. The current project focuses on increasing referrals to the Suicide Prevention 2.0 Clinical Telehealth (SP 2.0) initiative.

The investigators have recruited 4 sites for this non-randomized intervention project. Sites have agreed to participate in pre-implementation interviews to gather information regarding barriers and facilitators to use of the SP 2.0 initiative. Sites will then be provided with tailored feedback regarding interview findings and potential use of Academic Detailing and LEAP to address these. Sites may then select to receive either Academic Detailing and/or LEAP which will be provided by MIDAS QUERI. Primary outcome will be rate of SP 2.0 referral adjusted for pre-intervention rate.

ELIGIBILITY:
Inclusion Criteria:

Note- the investigators are recruiting clinics/medical centers - not individual patients. Prior to implementation, the investigators will work with sites to ensure they have met the preconditions necessary to begin sustained optimization of the EBP:

* 1) a team leader or champion
* 2) an identified department with service leadership buy-in and control over the processes/practices impacted by the implementation
* 3) readily accessible data to measure process and impact of the implementation and use of the EBP
* 4) availability of required resources

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul N Pfeiffer, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Jacob E Kurlander, MD MS MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Jeremy B. Sussman, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Site-level data that underlie results reported, after de-identification will be available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: For 36 months after article is published.
Access Criteria: Upon request by researchers who provide a methodologically sound proposal. Further details will be available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VA medical centers were recruited through Veterans Integrated Service Network (VISN) ICC calls and presentations to interested sites from November 2022 through May 2023. VISNs of interest were identified based on sites within that VISN having documented gaps in referring to the program.
Pre-assignment Details: 13 sites within VISNs of interest were approached directly. Following introductory presentations, 4 sites agreed to participate in the intervention arm. Four non-enrolled control sites were matched to the intervention arm sites based on size and baseline referral rates.
Units Other Than Participants: VA Medical Centers
Groups:
- Control: To examine the effect of engagement in quality improvement activity on referral to the SP2.0 program, we compared participating sites with similar non-participating sites. Four non-participating sites were selected as matched controls, one for each participating site. Control sites were matched to participating sites on number of suicide behavior events and prevalence of Suicide Prevention Telehealth Program consults submitted at baseline.
Period: Overall Study
Arm/Group | Intervention | Control
Started | NA; 4 VA Medical Centers (Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.) | NA; 4 VA Medical Centers (Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.)
Completed | NA; 4 VA Medical Centers (Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.) | NA; 4 VA Medical Centers (Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.)
Not Completed | NA; 0 VA Medical Centers | NA; 0 VA Medical Centers

BASELINE CHARACTERISTICS:
Population: The data came from a dashboard provided by an operational office and did not include demographics.
Units Other Than Participants: VA Medical Centers
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (VA Medical Centers) | 0 | 0 | 0
Age, Categorical — Population: Data on age was not collected nor was it available at the medical center level from our data source.
Sex: Female, Male — Population: Data on sex was not collected nor was it available at the medical center level from our data source.
Race/Ethnicity, Customized — Population: Data on race/ethnicity was not collected nor was it available at the medical center level from our data source.

OUTCOME MEASURES:

1. Primary Outcome: SP2Clin Metric
Description: The quarterly SP2Clin metric data is reported and available on a VA national dashboard. The SP2Clin metric is calculated by the number of suicide prevention telehealth consults submitted among those with a suicide behavior event.
Time Frame: Baseline to 12-months post-baseline
Population: Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.
Measure: Mean (Standard Deviation); unit: telehealth consults
Units Other Than Participants: VA Medical Centers
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (VA Medical Centers) | 4 | 4
telehealth consults | 22.6 (4.1) | 20.0 (3.8)
Statistical Analysis 1: Comparison: Intervention vs Control; We compared participating sites with similar non-participating sites. Four non-participating sites were selected as matched controls, one for each participating site. Control sites were matched to participating sites on number of suicide behavior events and prevalence of Suicide Prevention Telehealth Program consults submitted at baseline; Test type: Superiority — T-test to evaluate the effect of the intervention compared to control sites on reported suicide behavior events in the past 4 quarters that had an SP 2.0 Consult submitted; p = 0.5747, t-test, 2 sided; degrees of freedom = 6

2. Secondary Outcome: Change in Number of Consults to SP 2.0 Clinic
Description: Change in number of telehealth consults to the Suicide Prevention 2.0 Clinical Telehealth (SP 2.0) initiative.
Time Frame: Baseline to 12-months post-baseline
Population: Participants are not enrolled in this study. All enrollment and analysis were conducted at the VAMC level.
Measure: Mean (Standard Deviation); unit: telehealth consults
Units Other Than Participants: VA Medical Centers
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (VA Medical Centers) | 4 | 4
telehealth consults | 289.0 (171.3) | 256.0 (191.2)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — T-test to evaluate the effect of the intervention compared to control sites on referrals to the SP 2.0 Clinic; p = 0.8057, t-test, 2 sided; Degrees of freedom = 6

3. Other Pre Specified Outcome: Change in Quality Improvement Skills Application
Description: 16-item measure of change in quality improvement skills application. Values 1 to 4 where higher values indicate more frequent use of quality improvement skills.
Time Frame: Baseline to 12-months post-baseline
Population: This measure is only administered for those who participate in LEAP; this measure was not administered as no sites elected to participate in LEAP.
Units Other Than Participants: VA Medical Centers
Arm/Group | Intervention
Number analyzed (Participants) | NA
Number analyzed (VA Medical Centers) | 0

4. Other Pre Specified Outcome: Provider Satisfaction With Academic Detailing
Description: 7-items measuring satisfaction with Academic Detailing. Each response option uses a Likert-type scale with values 1 to 5 where higher values indicate higher satisfaction.
Time Frame: Post-first Academic Detailing session
Population: Participants were providers at participating sites who had received at least one AD session. AD satisfaction data was collected at the individual level; however, no demographic data was collected.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
Units on a scale | 4.75 (0.43)

5. Other Pre Specified Outcome: Change in Provider Satisfaction With LEAP
Description: 6-item measure of satisfaction with LEAP. Values 1 to 5 where higher values indicate higher satisfaction.
Time Frame: Baseline to 12-months post-baseline
Population: as for outcome 3
Units Other Than Participants: VA Medical Centers
Arm/Group | Intervention
Number analyzed (Participants) | NA
Number analyzed (VA Medical Centers) | 0

ADVERSE EVENTS:
Description: Adverse events were not monitored
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Site-level engagement in the intervention components was limited across sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT06011759/Prot_SAP_000.pdf